CLINICAL TRIAL: NCT03861780
Title: Pilot Evaluation of Two Test Materials With a Positive Control When Used as a Patient Preoperative Skin Preparation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Professional Disposables International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1810480-103
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Bacteria Microflora Reduction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Samples are blinded to the participant and technical team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Project X 26ml (Experimental): 3.15% w/v CHG (chlorhexidine gluconate) / 70% v/v IPA (isopropyl alcohol) contained within a saturated at use applicator. 26ml volume. Single use.
  Interventions: Drug: Project X 26ml
- Project X 5.1ml (Experimental): 3.15% w/v CHG (chlorhexidine gluconate) / 70% v/v IPA (isopropyl alcohol) contained within a saturated at use applicator. 5.1ml volume. Single use.
  Interventions: Drug: Project X 5.1ml
- Prevantics Maxi Swabstick (Active Comparator): 3.15% w/v CHG (chlorhexidine gluconate) / 70% v/v IPA (isopropyl alcohol). Swabstick. Single use.
  Interventions: Drug: Prevantics Maxi Swabstick

INTERVENTIONS:
Drug: Project X 26ml — Application of antiseptic drug to the inguinal and abdomen areas of the subjects
  Arms: Project X 26ml
Drug: Project X 5.1ml — Application of antiseptic drug to the inguinal and abdomen areas of the subjects
  Arms: Project X 5.1ml
Drug: Prevantics Maxi Swabstick — Application of antiseptic drug to the inguinal and abdomen areas of the subjects
  Arms: Prevantics Maxi Swabstick

SUMMARY:
Comparative Study of Antimicrobial Effectiveness Evaluation of 26ml Project X, 5.1ml Project X and Prevantics Maxi Swabstick following ASTM E1173 - Standard Test Method for Evaluation of Preoperative, Precatheterization, or Preinjection Skin Preparations, ASTM International, West Conshohocken, Pennsylvania, 2015

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, at least 18 years of age, and of any race.
* Subjects must be able to read and understand English.
* Subjects must have read and signed an Informed Consent Form, Authorization to Use and Disclose Protected Health Information Form, and List of Restricted Products prior to participating in the study, all located in the separate Informed Consent documents.
* Subjects must be in good general health and have no medical diagnosis of a physical condition, such as a current or recent severe illness, medicated or uncontrolled diabetes, hepatitis B, hepatitis C, an organ transplant, mitral valve prolapse with heart murmur, fibromyalgia, ulcerative colitis, Crohn's disease, an immunocompromised condition such as AIDS (or HIV positive), lupus, or medicated multiple sclerosis.
* Subjects will have test sites on the skin of the abdomen and/or inguinal free of injury and in good condition (no active skin rashes, excessive freckling, moles, scratches, breaks in the skin, etc.) and have no currently active skin diseases or skin conditions (for example, contact dermatitis, psoriasis or eczema) that may compromise subject safety or study integrity.
* Subjects must have skin within 6 inches of the test sites that is free of tattoos, dermatoses, abrasions, cuts, lesions or other skin disorders. Subjects with tattoos, scars, active skin rashes, or breaks in the skin of test sites, skin blemishes, such as dry scabs or warts, may be admitted at the discretion of the Principal Investigator, Subinvestigators, or Consulting Physicians.

Exclusion Criteria:

* Known allergies to vinyl, latex (rubber), alcohols, metals, tapes or adhesives, inks, sunscreens, deodorants, laundry detergents, topically applied fragrances, cleansers, or to common antibacterial agents found in soaps or lotions, particularly chlorhexidine gluconate or ethanol.
* Have experienced hives (raised welts) as a reaction to anything that contacted the skin.
* Use of systemic or topical antibiotic medications during the 14-day pre-test period through completion of testing on the single test day.
* Use of systemic or topical steroids, other than for contraception, hormone therapy, post-menopausal indications, during the 14-day pre-test period through completion of testing on the single test day. This includes steroid medications used to treat asthma. Note: topically applied hormonal steroids used for post-menopausal reasons must not get on the test sites.
* Any type of port (or portacath) or Peripherally Inserted Central Catheter (PICC).
* Pregnancy, plans to become pregnant or impregnate a sexual partner within the pre-test and test period of the study, or nursing a child. Female subjects must have a negative urine pregnancy test documented before treatment with test materials.
* Current participation or participation in a clinical study in the past 14 days.
* Any medical condition or use of any medications that, in the opinion of the Principal Investigator or consulting physicians, would preclude participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Collette Duley, Principal Investigator — BioScience Laboratories, Inc.
Locations (1):
- Bioscience Laboratories Inc, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 152 subjects were consented, randomized into the study, treated with test product and completed the study. Each subject is able to receive 2 test products (1 on each side of their body).
Groups:
- Project X 26ml: 3.15% w/v CHG / 70% v/v IPA contained within a saturated at use applicator. 26ml volume. Single use.
  Project X 26ml: Application of antiseptic drug to the inguinal and abdomen areas of the subjects
- Project X 5.1ml: 3.15% w/v CHG / 70% v/v IPA contained within a saturated at use applicator. 5.1ml volume. Single use.
  Project X 5.1ml: Application of antiseptic drug to the inguinal and abdomen areas of the subjects
- Prevantics Maxi Swabstick: 3.15% w/v CHG / 70% v/v IPA. Swabstick. Single use.
  Prevantics Maxi Swabstick: Application of antiseptic drug to the inguinal and abdomen areas of the subjects
Period: Overall Study
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Started | 51 | 50 | 51
Completed | 51 | 50 | 51
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick | Total
Number analyzed (Participants) | 51 | 50 | 51 | 152
Age, Continuous [Mean (Full Range); unit: years] | 42.1 [18 to 87] | 43.4 [18 to 87] | 44.7 [18 to 87] | 43.4 [18 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 28 | 78
  Male | 29 | 22 | 23 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 40 | 40 | 118
  Not Hispanic or Latino | 7 | 5 | 4 | 16
  Unknown or Not Reported | 6 | 5 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Bacterial Microflora on the Inguinal Area
Description: Bacterial microflora (log10) will be measured via cup scrub method administration of the intervention
Time Frame: 30 seconds
Population: The overall number of participants analyzed represents the modified intent to treat (mITT) data set. The Participant Flow was is based on the intent to treat (ITT) dataset. Additionally, each subject is able to receive 2 test products (1 on each side of their body).
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 30 | 29 | 27
Number analyzed (evaluable sites) | 59 | 58 | 53
log10 CFU | -3.7 (1.4) | -3.1 (1.3) | -3.5 (1.4)

2. Primary Outcome: Change in Bacterial Microflora on the Inguinal Area
Description: Bacterial microflora (log10) will be measured via cup scrub method administration of the intervention
Time Frame: 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 29 | 29 | 27
Number analyzed (evaluable sites) | 58 | 58 | 53
log10 CFU | -3.5 (1.2) | -3.2 (1.5) | -3.3 (1.6)

3. Primary Outcome: Change in Bacterial Microflora on the Inguinal Area
Description: Bacterial microflora (log10) will be measured via cup scrub method administration of the intervention
Time Frame: 6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 30 | 29 | 27
Number analyzed (evaluable sites) | 59 | 58 | 53
log10 CFU | -3.8 (1.3) | -3.6 (1.5) | -3.4 (1.4)

4. Primary Outcome: Change in Bacterial Microflora on the Abdomen Area
Description: Bacterial microflora (log10) will be measured via cup scrub method administration of the intervention
Time Frame: 30 seconds
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 25 | 29 | 29
Number analyzed (evaluable sites) | 50 | 57 | 57
log10 CFU | -3.2 (1.1) | -2.9 (1.1) | -2.8 (1.1)

5. Primary Outcome: Change in Bacterial Microflora on the Abdomen Area
Description: Bacterial microflora (log10) will be measured via cup scrub method administration of the intervention
Time Frame: 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 25 | 29 | 29
Number analyzed (evaluable sites) | 50 | 57 | 57
log10 CFU | -3.0 (1.2) | -2.9 (1.1) | -2.9 (1.0)

6. Primary Outcome: Change in Bacterial Microflora on the Abdomen Area
Description: Bacterial microflora (log10) will be measured via cup scrub method administration of the intervention
Time Frame: 6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 26 | 29 | 29
Number analyzed (evaluable sites) | 51 | 58 | 57
log10 CFU | -2.9 (1.0) | -3.0 (1.0) | -2.7 (1.0)

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Project X 26 mL: 3.15% w/v CHG (chlorhexidine gluconate) / 70% v/v IPA (isopropyl alcohol) contained within a saturated at use applicator. 26ml volume. Single use.
  Project X 26ml: Application of antiseptic drug to the inguinal and abdomen areas of the subjects
- Project X 5.1 mL: 3.15% w/v CHG (chlorhexidine gluconate) / 70% v/v IPA (isopropyl alcohol) contained within a saturated at use applicator. 5.1 ml volume. Single use.
  Project X 5.1 ml: Application of antiseptic drug to the inguinal and abdomen areas of the subjects
- Prevantics Maxi Swabstick: 3.15% w/v CHG (chlorhexidine gluconate) / 70% v/v IPA (isopropyl alcohol) Swabstick. Single use.
  Application of antiseptic drug to inguinal and abdomen areas of the subjects
Arm/Group | Project X 26 mL | Project X 5.1 mL | Prevantics Maxi Swabstick
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 1/51 | 0/50 | 0/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Project X 26 mL (N=51) | Project X 5.1 mL (N=50) | Prevantics Maxi Swabstick (N=51)
Treatment Related AE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Study-related non-serious, Treatment Emergent AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT03861780/Prot_SAP_000.pdf